CLINICAL TRIAL: NCT00091442
Title: A Randomized Controlled Study of Docetaxel Monotherapy or Docetaxel and DOXIL for the Treatment of Advanced Breast Cancer
Brief Title: A Study of Docetaxel Monotherapy or DOXIL and Docetaxel in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004120; DOXILBCA3001 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); NCT00343538 (obsolete NCT alias)
Record Dates: First submitted 2004-09-08; First posted 2004-09-13 (Estimated); Results first posted 2012-10-02 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Advanced breast cancer; Breast Tumors; Cancer of Breast; Human Mammary Carcinoma; Mammary Neoplasms, Human; DOXIL; Docetaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DOXIL and docetaxel combination therapy (Experimental): DOXIL and docetaxel combination therapy: DOXIL 30 mg/m2 solution administered by intravenous infusion, followed by docetaxel 60 mg/m2 administration by intravenous infusion over 1 hour on Day 1 of every 21-day cycle.
  Interventions: Drug: Docetaxel; Drug: DOXIL
- Docetaxel monotherapy (Active Comparator): Docetaxel monotherapy: Docetaxel 75 mg/m2 solution administered by intravenous infusion over 1 hour on Day 1 of every 21-day cycle
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Docetaxel monotherapy: docetaxel 75 mg/m2 solution administered by intravenous infusion over 1 hour on Day 1 of every 21-day cycle. DOXIL in combination with docetaxel: docetaxel 60 mg/m2 solution administered by intravenous infusion over 1 hour on Day 1 of every 21-day cycle
Drug: DOXIL — DOXIL 30 mg/m2 solution administered by intravenous infusion over 1 hour on Day 1 of every 21-day cycle.
  Other Names: DOXIL in combination with Docataxel
  Arms: DOXIL and docetaxel combination therapy

SUMMARY:
The purpose of the study is to evaluate whether the time to progression for the DOXIL and docetaxel combination therapy group was superior to that of the group treated with docetaxel monotherapy in participants with advanced breast cancer.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by a random order), active control (study medication will be compared with available standard care of treatment), parallel-group (each treatment group will be treated simultaneously at the same time and each participant only receives one treatment regimen as assigned), open-label (both the investigator and the participant know the intervention received by the participant), multicenter study designed to determine if women with locally advanced or metastatic breast cancer, who were previously treated with prior anthracycline therapy in the neoadjuvant (administration of treatment before surgery) or adjuvant setting (administration of treatment after surgery), and who also had a disease-free interval of at least 12 months since the end of their last cytotoxic therapy, would benefit from the addition of DOXIL to docetaxel therapy. Approximately 751 participants will be randomly assigned to either receive docetaxel monotherapy or DOXIL in combination with docetaxel therapy. Treatment is to continue until disease progression or the occurrence of unacceptable treatment related toxicity. Safety evaluations will include assessments of adverse events which will be recorded from the first study related procedure until 30 days after the last dose of medication; clinical laboratory tests and tests for cardiac function (multiple gated acquisition scan/echocardiogram and electrocardiogram) which will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Females with locally advanced or metastatic breast cancer who received prior anthracycline therapy in the neoadjuvant or adjuvant setting, and had at least a 12-month disease-free interval since the end of their last cytotoxic therapy, were eligible for the study
* Participants who received prior hormonal therapy, or no more than 1 cytotoxic chemotherapy regimen (anthracyclines, taxanes, or antitubulin agents were not permitted), or both for advanced disease
* Participants with normal cardiac function, as evidenced by a normal left ventricular ejection fraction

Exclusion Criteria:

* More than 1 prior cytotoxic chemotherapy regimen for advanced breast cancer
* Treatment of advanced breast cancer with an anthracycline, paclitaxel, docetaxel, vinorelbine, or vinblastine (prior treatment of advanced breast cancer with 1 regimen that included alkylating agents or antimetabolite agents was acceptable)
* Less than 2 months since the last dose of trastuzumab
* Less than 3 weeks since last dose of tamoxifen or fulvestrant, or less than 1 week since the last dose of other hormonal therapy
* Radiation to areas of disease within 30 days before study enrollment
* History of New York Heart Association Class II or greater cardiac disease or other clinical evidence of congestive heart failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2004-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (147):
- United States (30):
  - Hoover, Alabama
  - Fountain Valley, California
  - Long Beach, California
  - Los Angeles, California
  - Palm Springs, California
  - Newark, Delaware
  - Lakeland, Florida
  - Fort Gordon, Georgia
  - Centralia, Illinois
  - Joliet, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Lafayette, Louisiana
  - Baltimore, Maryland
  - Jackson, Mississippi
  - Las Vegas, Nevada
  - Newark, New Jersey
  - Albuquerque, New Mexico
  - Cooperstown, New York
  - New York, New York
  - The Bronx, New York
  - Gastonia, North Carolina
  - Philadelphia, Pennsylvania
  - Upland, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - North Charleston, South Carolina
  - Fort Worth, Texas
  - Pasadena, Texas
- Bulgaria (5):
  - Plovdiv
  - Shumen
  - Sofia
  - Stara Zagora
  - Varna
- Tartu, Estonia
- France (2):
  - Rabat-les-Trois-Seigneurs
  - Tunis
- Hungary (5):
  - Budapest
  - Debrecen
  - Szeged
  - Székesfehérvár
  - Zalaegerszeg
- Israel (5):
  - Ashkelon
  - Haifa
  - Jerusalem
  - Ramat Gan
  - Tel Aviv
- Riga, Latvia
- Lithuania (2):
  - Kaunas
  - Vilnius
- Netherlands (4):
  - Arnhem
  - Capelle aan den IJssel
  - Roosendaal
  - The Hague
- Poland (14):
  - Bialystok
  - Bydgoszcz
  - Bytom
  - Gdansk
  - Gdynia
  - Gliwice
  - Kielce
  - Koszalin
  - Krakow
  - Lodz
  - Lublin
  - Olsztyn
  - Poznan
  - Warsaw
- Portugal (2):
  - Coimbra
  - Matosinhos Municipality
- Romania (7):
  - Bacau
  - Bucharest
  - Cluj-Napoca
  - Hunedoara
  - Iași
  - Onești
  - Timișoara
- Russia (36):
  - Arkhangelsk
  - Balashikha
  - Barnaul
  - Chelyabinsk
  - Engels Saratov Region
  - Irkutsk
  - Ivanovo
  - Izhevsk
  - Kazan'
  - Krasnodar
  - Leningrad Region
  - Lipetsk
  - Moscow
  - Moscow Region
  - Murmansk
  - Nizhny Novgorod
  - Novosibirsk
  - Obninsk
  - Omsk
  - Oryol
  - Petrozavodsk
  - Pyatigorsk
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Samara
  - Smolensk
  - Stavropol
  - Tomsk
  - Tver'
  - Ulyanovsk
  - Vladimir
  - Volgograd
  - Voronezh
  - Yaroslavl
  - Yekaterinburg
- Serbia (3):
  - Belgrade
  - Kamenitz
  - Niš
- South Africa (7):
  - Cape Town
  - Johannesburg
  - Kimberley
  - Parktown
  - Port Elizabeth
  - Pretoria
  - Pretoria Gauteng
- Spain (5):
  - Bilbao Vizcaya
  - Lleida
  - Madrid
  - Santander
  - Seville
- Ukraine (14):
  - Cherkassy
  - Chernivtsi
  - Dnipro
  - Donetsk
  - Kharkiv
  - Kiev
  - Luhansk
  - Lutsk
  - Odesa
  - Poltava
  - Simferopol
  - Uzhhorod
  - Vinnitsa
  - Zhytomyr
- United Kingdom (4):
  - Huddersfield
  - Manchester
  - Nottingham
  - Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 751 participants were enrolled and randomized at 143 sites in 19 countries.
Pre-assignment Details: 751 participants were randomly assigned to 2 treatment groups (Docetaxel: 373 ; DOXIL+docetaxel: 378). 750 participants received treatment (Docetaxel: 373; DOXIL+docetaxel: 377). 1 participant in DOXIL+docetaxel treatment group did not receive treatment.
Groups:
- Docetaxel: Docetaxel monotherapy: Docetaxel 75 mg/m2 solution administered by intravenous infusion over 1 hour on Day 1 of every 21-day cycle.
- DOXIL+Docetaxel: DOXIL and docetaxel combination: DOXIL 30 mg/m2 solution administered by intravenous infusion, followed by docetaxel 60 mg/m2 administration by intravenous infusion over 1 hour on Day 1 of every 21-day cycle.
Period: Overall Study
Arm/Group | Docetaxel | DOXIL+Docetaxel
Started | 373 | 378
Completed | 4 (Indicates number of participants on study treatment at time of the primary objective) | 5 (Indicates number of participants on study treatment at time of the primary objective)
Not Completed | 369 | 373
Not completed — Progressive Disease | 220 | 189
Not completed — Physician Decision | 61 | 58
Not completed — Withdrawal by Subject | 38 | 46
Not completed — Adverse Event | 29 | 48
Not completed — 2cycles therapy beyond Complete response | 9 | 16
Not completed — Death | 9 | 7
Not completed — Lost to Follow-up | 1 | 3
Not completed — Other | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel | DOXIL+Docetaxel | Total
Number analyzed (Participants) | 373 | 378 | 751
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (9.23) | 52.8 (9.17) | 52.4 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 373 | 378 | 751
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Overall Survival
Description: Time interval in months between the date of randomization and the participant's death from any cause.
Time Frame: From the date of randomization until the participant's death from any cause, as assessed until approximately 485 death events were observed which is assessed approximately 25 months after the last patient was enrolled
Population: Intent to Treat: If the date of death was unknown, the data were censored at the date that the participant was last known to have been alive.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | DOXIL+Docetaxel
Number analyzed (Participants) | 373 | 378
Months | 20.7 [18.3 to 26.3] | 20.4 [19.0 to 23.1]
Statistical Analysis 1: Comparison: Docetaxel vs DOXIL+Docetaxel; Null Hypothesis: Designed to detect an improvement in median survival from 15 months to 19.5 months with 80% power; Test type: Superiority or Other; p = 0.5988, Log Rank — Not adjusted for multiple comparison; Hazard Ratio (HR) = 1.06, 95% CI [0.86 to 1.3]

2. Secondary Outcome: Response Rate: Number of Participants in the Evaluable Population Who Achieved a Complete Response (CR) or Partial Response (PR)
Description: Number of participants in the evaluable population who achieved a CR or PR as per Response Evaluation Criteria In Solid Tumors (RECIST) criteria. CR: Disappearance of all target lesions and PR: at least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD. Response was assessed by Computed Tomography (CT)/Magnetic Resonance Imaging (MRI).
Time Frame: Up to 30 to 42 days after last dose of study medication
Population: Evaluable population: Included all randomized participants who received at least 1 dose of study medication (DOXIL or docetaxel), and who had at least 1 postbaseline tumor assessment.
Measure: Number; unit: Participants
Arm/Group | Docetaxel | DOXIL+Docetaxel
Number analyzed (Participants) | 364 | 370
Participants | 95 | 129
Statistical Analysis 1: Comparison: Docetaxel vs DOXIL+Docetaxel; Null hypothesis - no difference in response rate between the two treatment groups; Test type: Superiority or Other; p = 0.0085, Cochran-Mantel-Haenszel — Not adjusted for multiple comparison

3. Primary Outcome: Time to Progression
Description: Time interval in months between the date of randomization and the date of disease progression or death due to progression, whichever occurred first.
Time Frame: From date of randomization until date of disease progression or death, whichever occurred first, until approximately 485 events of disease progression or death were observed, as assessed approximately 15 months after the last patient was enrolled
Population: Intent to Treat: For patients who were progression free at the time of data cutoff, data were censored for time to progression at the time of their last tumor assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | DOXIL+Docetaxel
Number analyzed (Participants) | 373 | 378
Months | 7.0 [5.9 to 7.7] | 9.8 [8.1 to 10.5]
Statistical Analysis 1: Comparison: Docetaxel vs DOXIL+Docetaxel; Null hypothersis - no difference in Time to Progression (TTP) between the two treatment groups. Designed to detect an improvement in median TTP from 6 months to 7.8 months with 80% power, assuming exponential survival distribution; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.65, 95% CI [0.55 to 0.77]

ADVERSE EVENTS:
Time Frame: From first dose of study medication until 30 days after the last dose of study medication.
Description: 751 participants were randomly assigned to 2 treatment groups (Docetaxel: 373 ; DOXIL+docetaxel: 378). 750 participants received treatment (Docetaxel: 373; DOXIL+docetaxel: 377). 1 participant in DOXIL+docetaxel treatment group did not receive treatment.
Arm/Group | Docetaxel | DOXIL+Docetaxel
Serious Adverse Events (participants affected / at risk) | 59/373 | 69/377
Other Adverse Events (participants affected / at risk) | 340/373 | 359/377
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=373) | DOXIL+Docetaxel (N=377)
Neutropenia (Blood and lymphatic system disorders) | 14 | 17
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 10
Leukopenia (Blood and lymphatic system disorders) | 1 | 4
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 12
Neutropenic sepsis (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Catheter site cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Pulpitis dental (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Vulvitis (Infections and infestations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 3 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 6
Asthenia (General disorders) | 1 | 3
Infusion related reaction (General disorders) | 0 | 2
Death (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
cardiac failure (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Cardiac disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1
Heachache (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 0 | 2
Brain stem syndrome (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 7
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Superior vena caval occlusion (Vascular disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Alanine aminotransferease increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Surgery (Surgical and medical procedures) | 0 | 1
Uterine dilation and curettage (Surgical and medical procedures) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=373) | DOXIL+Docetaxel (N=377)
Anaemia (Blood and lymphatic system disorders) | 62 | 75
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 19
Leukopenia (Blood and lymphatic system disorders) | 99 | 126
Neutropenia (Blood and lymphatic system disorders) | 241 | 244
Tachycardia (Cardiac disorders) | 14 | 21
Constipation (Gastrointestinal disorders) | 18 | 13
Diarrhoea (Gastrointestinal disorders) | 42 | 56
Mucositis/stomatitis (Gastrointestinal disorders) | 53 | 195
Nausea (Gastrointestinal disorders) | 80 | 105
Vomiting (Gastrointestinal disorders) | 35 | 38
Asthenia (General disorders) | 72 | 110
Fatigue (General disorders) | 56 | 78
Oedema peripheral (General disorders) | 34 | 17
Pyrexia (General disorders) | 31 | 59
Respiratory tract infection (Infections and infestations) | 12 | 21
Alanine aminotransferase increased (Investigations) | 29 | 31
Aspartate aminotransferase increased (Investigations) | 31 | 26
Weight decreased (Investigations) | 6 | 18
Anorexia (Metabolism and nutrition disorders) | 21 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 26
Bone pain (Musculoskeletal and connective tissue disorders) | 26 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 33 | 32
Dizziness (Nervous system disorders) | 12 | 18
Dysgeusia (Nervous system disorders) | 22 | 10
Headache (Nervous system disorders) | 21 | 39
Peripheral neuropathy (Nervous system disorders) | 68 | 78
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 | 29
Alopecia (Skin and subcutaneous tissue disorders) | 169 | 181
Erythema (Skin and subcutaneous tissue disorders) | 6 | 17
Nail disorder (Skin and subcutaneous tissue disorders) | 26 | 37
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 229

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission. Expedited reviews will be arranged if needed. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application. The sponsor will not mandate modifications to scientific content and does not have the right to suppress information.